CLINICAL TRIAL: NCT02413047
Title: A Pilot Study to Evaluate if Response to Infliximab or Adalimumab May be Regained With the Addition of an Immunomodulator
Brief Title: Evaluate if Response to Infliximab or Adalimumab May be Regained With an Immunomodulator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: physician decision to stop study early due to low enrollment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Matthew Bohm, Assistant Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1502834262
Record Dates: First submitted 2015-03-06; First posted 2015-04-09 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Azathioprine; Mercaptopurine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunomodulator (Experimental): Azathioprine, 6 mercaptopurine or methotrexate.
  Interventions: Drug: Azathioprine; Drug: 6 mercaptopurine; Drug: Methotrexate

INTERVENTIONS:
Drug: Azathioprine — Medication will be given in pill form to patients to take daily as long as the patient has not been intolerant to it in the past.
  Other Names: Imuran
Drug: 6 mercaptopurine — Medication will be given in pill form to patients to take daily as long as the patient has not been intolerant to it in the past as an alternative to imuran
Drug: Methotrexate — Medication will be given in subcutaneous injection form once a week if the patient cannot take imuran or 6 mercaptopurine.

SUMMARY:
The immunogenicity of anti-tumor necrosis factor alpha (anti-TNF) therapy in inflammatory bowel disease (IBD) is an important cause of loss of response to therapy that may lead to escalation of dose or discontinuation of therapy. Antibodies may develop to infliximab (ATI) or to adalimumab (ATA) and cause this loss of response, also known as a secondary loss of response. An alternative approach is the addition of immunomodulator (IM) therapy to counteract the antibody response and regain efficacy of the biologic medication. The investigators' goal is to treat patients' who have lost response to adalimumab or infliximab with an immunomodulator with the goal of eliminating the circulating antibodies to the anti-TNF and restoring efficacy.

DETAILED DESCRIPTION:
The immunogenicity of anti-tumor necrosis factor alpha (anti-TNF) therapy in inflammatory bowel disease (IBD) is an important cause of loss of response to therapy that may lead to escalation of dose or discontinuation of therapy. Antibodies may develop to infliximab (ATI) or to adalimumab (ATA) and cause this loss of response, also known as a secondary loss of response. In an attempt to overcome these antibodies, dose escalation can be accomplished either by increasing the dose or shortening the interval between doses. The ability of dose escalation to overcome loss of response due to the presence of ATI or ATA remains controversial. Escalation of dose increases the cost of therapy substantially. If the decision is made to discontinue therapy after a secondary loss of response, a clinician may choose to switch to an alternate anti-TNF therapy of which there are currently only four. Loss of response to one agent predicts a lesser response to other anti-TNF agents and with a limited number of therapeutic options the goal should be to optimize therapy rather than to discontinue therapy.

An alternative approach is the addition of immunomodulator (IM) therapy to counteract the antibody response and regain efficacy of the biologic medication. Three such IMs known to be effective in the treatment of IBD are azathioprine (AZA), 6-mercaptopurine (6MP) and methotrexate (MTX). The SONIC trial showed that patients on infliximab and azathioprine only developed antibodies at 4% of the time as opposed to those on infliximab monotherapy who formed ATI at 13%. The same principal was shown during the COMMIT trial in which patients on infliximab alone had ATI at a rate of 20% versus 4% on methotrexate plus infliximab. Ben-Horin et al. reported five patients treated initially with infliximab monotherapy whom had secondary loss of response based on clinical symptoms. These patients had ATI and all had undetectable troughs of infliximab. In all five patients ATI became undetectable, an adequate trough level was restored and the patients regained clinical response with the addition of an immunomodulator. Combination therapy with azathioprine and infliximab has led to a higher percentage of patients in steroid free remission than either drug alone. Our goal is to treat patients' who have lost response to adalimumab or infliximab with an immunomodulator with the goal of eliminating the circulating antibodies to the anti-TNF and restoring efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease who on are stable doses of infliximab or adalimumab for at least 3 months who experience a secondary loss of response to the medication based on clinical symptoms.
* Presence of at least one objective marker of active disease: active disease based on endoscopy, elevated fecal calprotectin or serologic markers of inflammation (C-reactive protein or sedimentation rate).
* Crohn's patients have a Harvey Bradshaw index >5
* Ulcerative colitis patients have a Ulcerative Colitis Clinical Score > 5
* Have an undetectable or inadequate trough level of infliximab or adalimumab and detectable ATI or ADA.
* Oral corticosteroid therapy is allowed. (prednisone at a stable dose ≤30 mg/day, budesonide at a stable dose ≤9 mg/day, or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to enrollment if corticosteroids have recently been initiated

Exclusion Criteria:

* Previous noncompliant with medications
* < 18 years of age or >80 years of age.
* Congestive heart failure
* Abnormal liver tests alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2 × the upper limit of normal (ULN) or leucopenia WBC count <3 × 109/L
* Pregnant or planning on becoming pregnant.
* Active tuberculosis or hepatitis B infection
* Any cancer within the past 5 years. (Exception non-melanomatous skin cancer.)
* Receiving any immunomodulator therapy within the past 3 months
* Evidence of or treatment for C. difficile infection within 60 days or other intestinal pathogen within 30 days prior to enrollment
* Clinically significant extra-intestinal infection (e.g., pneumonia, pyelonephritis) within 30 days of the initial screening visit
* Any live vaccinations within 30 days prior to study drug administration except for the influenza vaccine
* Any identified congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation)
* Any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise patient safety
* Unable to give own informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bohm, DO, Principal Investigator — IndianaU IRB
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data was analyzed

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immunomodulator
Started | 3
Participants on Infliximab | 2
Participants on Adalimumab | 1
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Not enough study participants enrolled for data analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
Duration of Disease [Mean (Full Range); unit: years] | 16.66666667 [4 to 40]
White Blood Cell Count (WBC) [Mean (Full Range); unit: x 10^3 cells/mm^3] | 6.566666667 [6.2 to 7.0]
Hemoglobin [Mean (Full Range); unit: gm/dL] | 13.63 [12.6 to 14.5]
Platelet Count [Mean (Full Range); unit: x 10^3 cells/mm^3] | 256.00 [237 to 292]
Aspartate Aminotransferase [Mean (Full Range); unit: units/L] | 21.00 [16 to 30]
ALT [Mean (Full Range); unit: units/L] | 23.67 [13 to 42]
Bilirubin [Mean (Full Range); unit: mg/dL] | 0.67 [0.60 to 0.70]
Albumin [Mean (Full Range); unit: gm/dL] | 4.37 [4.10 to 4.60]
Alkaline Phosphatase [Mean (Full Range); unit: units/L] | 93.33 [66 to 126]
Above-Normal C-Reactive Protein [Number; unit: mg/dL] — 'Normal" c-reactive protein levels are resulted as <0.5mg/dL Population: "Normal" c-reactive protein levels are resulted from the laboratory as '<0.5mg/dL'. Therefore, only levels higher than 0.5mg/dL will be reported.
  mg/dL
    number analyzed (Participants) | 1
    (all) | 2.0
Erythrocyte Sedimentation Rate [Mean (Full Range); unit: mm/hr] | 23.67 [15 to 34]
Calprotectin [Mean (Full Range); unit: mCg/gm] | 331.50 [232 to 431]
Simple Endoscopic Score for Crohn's Disease [Mean (Full Range); unit: points] — 0-2 = remission 3-6 = mild endoscopic activity 7-15 = moderate endoscopic activity >15 = severe endoscopic activity
  points | 6.67 [6.00 to 8.00]
Harvey Bradshaw Index (HBI) Score [Mean (Full Range); unit: points] — <5 = Remission 5-7 = mild activity 8-16 = moderate activity >16 = severe activity
  points | 4.67 [3 to 6]
Short Inflammatory Bowel Disease Questionnaire [Mean (Full Range); unit: points] — SIBDQ measure the quality of life in patients with IBD. Each question is graded from 1-7. outcomes vary with '32' (very poor quality of life) to 224 (perfect quality of life. Patients in systematic remission typically have a score of 170 or greater. An increase of 16-32 points constitutes clinically meaningful improvement.
  points | 46.00 [28 to 56]
Serum Infliximab concentration [Number; unit: ug/mL] — Trough Level: lowest level of drug detected in subjected prior to next dose. Population: Only 2 subjects of 3 subjects were on infliximab for the study. 1 of the 2 subjects had a undetectable trough level (<1) and the other subject level was 6.3.
  ug/mL
    number analyzed (Participants) | 1
    (all) | 6.3
Antibodies to Infliximab concentration [Mean (Full Range); unit: units/mL] — Population: 2 of the 3 subjects were on infliximab
  units/mL
    number analyzed (Participants) | 2
    (all) | 20.70 [18.5 to 22.9]
Serum Adalimumab concentration [Number; unit: ug/mL] — Trough level: lowest level of drug detected in subject prior to next dose Population: 1 of the 3 subjects were on adalimumab
  ug/mL
    number analyzed (Participants) | 1
    (all) | 2
Antibodies to Adalimumab concentration [Number; unit: units/mL] — Population: 1 of 3 subjects on Adalimumab
  units/mL
    number analyzed (Participants) | 1
    (all) | 2.8

OUTCOME MEASURES:

1. Primary Outcome: Harvey Bradshaw Index HBI: Decrease >3 Points or Remission Score<5
Description: The Harvey-Bradshaw index (HBI) is a simplified version of the CDAI to foster a systematic collection of clinical data related to Crohn's disease.
  The index considers five parameters, exclusively clinical; patient well-being, abdominal pain, number of liquid or soft stools, abdominal mass, and complications.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

2. Primary Outcome: Therapeutic Trough Level for Infliximab is Defined as >3 and as > 5 for Adalimumab.
Description: Trough level is the lowest level of drug detected in a subject prior to next dose of medication
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

3. Primary Outcome: Ulcerative Colitis Clinical Score UCCS Decrease >3 Points or Remission Score <3
Description: UCCS is the ulcerative colitis clinical score which is based on disease activity. The score is based on bowel movements, blood in stool, overall well being, and global assessment.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

4. Primary Outcome: Change Inflammatory Bowel Disease Questionnaire SIBDQ
Description: SIBDQ is the short inflammatory bowel disease questionnaire which is a health-related quality of life tool measuring physical, social, and emotional status.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

5. Primary Outcome: Eliminate Antibodies: Threshold Levels for ATI is < 3.1and is < 1.7 for ADA.
Description: unwanted immunogenicity is an immune response by an organism against a therapeutic antigen. This reaction leads to production of anti-drug antibodies inactivating the therapeutic effects of the treatment.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

6. Secondary Outcome: Improvement or Normalization of Mayo Endoscopy Score for UC Patients
Description: Mayo endoscopy score is scoring completed during the endoscopy to evaluate disease activity. Scoring is based on stool frequency, rectal bleeding, mucosal appearance at endoscopy, and physician rating of disease activity
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

7. Secondary Outcome: Improvement or Normalization of C-reactive Protein, Sedimentation Rate and Fecal Calprotectin
Description: c-reactive protein, sedimentation rate, and fecal calprotectin were collected to monitor the level of inflammation in the subject. Improvement was determined if inflammation level was reduced.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

8. Secondary Outcome: Improvement or Normalization of the Simple Endoscopic Score-Crohn's Disease (SES-CD)
Description: SESCD is the simple endoscopic score for crohn's disease patients scored during endoscopy. The scoring is based on appearance of ulcers/sizing, % of ulcerative surface, % of affected surface, and if there were any narrowings or strictures found.
Time Frame: 4 months
Population: Not enough subjects for analysis
Arm/Group | Immunomodulator
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Enrollment to 16 weeks
Arm/Group | Immunomodulator
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The study terminated early due to low subject enrollment. Since only 3 patients were enrolled, study analysis was not possible for measurable outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT02413047/Prot_SAP_000.pdf